CLINICAL TRIAL: NCT05304325
Title: Evaluation of Adipose Tissue Pre and Post Bariatric Surgery
Brief Title: Adipose Tissue Pre and Post Bariatric Surgery
Acronym: ETAPP
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Rémi Rabasa-Lhoret, Full professor, Institut de Recherches Cliniques de Montreal
Other Study IDs: 2011-22
Record Dates: First submitted 2022-03-14; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Obesity
Keywords: Bariatric surgery; Persistant organic pollutants; Type 2 diabetes
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery; Blood Specimen Collection; Blood Pressure; Body Composition; Basal Metabolism; Eating

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Obese with type 2 diabetes
  Interventions: Procedure: Bariatric surgery; Other: Blood sampling; Other: Blood pressure; Other: Anthropometric measurements; Other: Body composition; Other: Resting metabolic rate; Other: Food intake; Procedure: Adipose tissue biopsy
- Obese insulin-sensitive
  Interventions: Procedure: Bariatric surgery; Other: Blood sampling; Other: Blood pressure; Other: Anthropometric measurements; Other: Body composition; Other: Resting metabolic rate; Other: Food intake; Procedure: Adipose tissue biopsy
- Obese insulin-resistant
  Interventions: Procedure: Bariatric surgery; Other: Blood sampling; Other: Blood pressure; Other: Anthropometric measurements; Other: Body composition; Other: Resting metabolic rate; Other: Food intake; Procedure: Adipose tissue biopsy

INTERVENTIONS:
Procedure: Bariatric surgery — Sleeve gastrectomy
Other: Blood sampling — Blood samples will be collected to measure glucose, insulin, albumin, uric acid, HbA1c, lipids, hepatic enzymes, TSH, hs-CRP, complete blood cell counts and persistant organic pollutants
Other: Blood pressure — Systolic and diastolic blood pressure will be measured.
Other: Anthropometric measurements — Body weight, height and waist circumference will be measured.
Other: Body composition — Body composition will be evaluated by dual-energy X-ray absorptiometry.
Other: Resting metabolic rate — Resting metabolic rate will be measured by indirect calorimetry.
Other: Food intake — Food intake, energy intake and food quality will be evaluated using the food frequence questionnaire.
Procedure: Adipose tissue biopsy — A sample of 3-5g of adipose tissue will be collected under local anesthesia by needle aspiration in the periumbilical region.

SUMMARY:
Published data suggest that inflammation and fibrosis of adipose tissue could be factors favoring the development of insulin resistance in obese individuals and that a decrease in the activity of the AMP-activity kinase protein (AMPK) could lead to these dysfunctions. However, very few data are available in humans.

There is also growing interest in persistent organic pollutants (POPs) as a cardiometabolic and type 2 diabetes (T2D) risk factor. There is some evidence to suggest that POPs directly contribute to lipid metabolism dysfunction and insulin resistance. Additionally, POPs are stocked in adipose tissue. The accumulation of POPs in adipose tissue therefore limits their bioavailability to other organs, thus reducing their systemic toxicity. It has been observed that a large amplitude weight loss leads to a significant increase in POPs in the blood.

The goal of this project is to identify adipose tissue factors/dysfunctions that contribute to insulin resistance and type 2 diabetes associated with obesity in humans and thus raise avenues for screening and treatment of these metabolic complications. More specifically, the objectives are:

* To study the relationship between AMPK, fibrosis and inflammation of adipose tissue and their role in the development of insulin resistance and T2D associated with obesity;
* To examine the relationship between POPs and the cardiometabolic profile.

ELIGIBILITY:
Inclusion Criteria:

1. Awaiting bariatric surgery
2. BMI ≥ 35 kg/m2 without cardiometabolic complications or ≥ 30 kg/m2 if presence of type 2 diabetes or hypertension
3. ≥ 18 years old
4. Non smoker
5. Sedentary (less than 3 hours of regular physical activity per week)

Exclusion Criteria:

1. Type 1 diabetes
2. Acute event in the last 3 months (myocardial infarction, cerebrovascular hemorrhage or transient cerebral ischemia, unstable angina, peripheral vascular disease, revascularization or angioplasty, recent hospitalization for more than 4 days)
3. Infection in the last month (fever, antibiotics treatment)
4. Cancer in the last 3 years
5. Chronic inflammatory disease
6. Pharmacologic treatment (any medication affecting glucose metabolism (except those for diabetes), hypotensive medication unless stable dose for at least 1 month, lipid-lowering medication unless stable dose for at least 1 month)
7. Uncontrolled disease of pituitary or thyroid gland
8. Bleeding disorders
9. Alcohol or drug abuses
10. Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be composed of obese individuals with type 2 diabetes, insulin-sensitive obese individuals and insulin-resistant obese individuals, all awaiting bariatric surgery.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2012-04-25 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Adipose tissue fibrosis using qRT-PCR, immunoblotting, histochemistry and immunohistochemistry | Before bariatric surgery
Adipose tissue fibrosis using qRT-PCR, immunoblotting, histochemistry and immunohistochemistry | 6 months after bariatric surgery

SECONDARY OUTCOMES:
Calory intake | Before bariatric surgery
Calory intake | 3 months after bariatric surgery
Calory intake | 6 months after bariatric surgery
Food quality using the Food Frequency Questionnaire | Before bariatric surgery
Food quality using the Food Frequency Questionnaire | 3 months after bariatric surgery
Food quality using the Food Frequency Questionnaire | 6 months after bariatric surgery
Persistant organic pollutants measured by high-resolution chromatography combined with high-resolution mass spectrometry | Before bariatric surgery
Persistant organic pollutants measured by high-resolution chromatography combined with high-resolution mass spectrometry | 3 months after bariatric surgery
Persistant organic pollutants measured by high-resolution chromatography combined with high-resolution mass spectrometry | 6 months after bariatric surgery
AMP-activated protein kinase | Before bariatric surgery
AMP-activated protein kinase | 3 months after bariatric surgery
AMP-activated protein kinase | 6 months after bariatric surgery
Inflammation in adipose tissue using qRT-PCR, immunoblotting and immunohistochemistry | Before bariatric surgery
Inflammation in adipose tissue using qRT-PCR, immunoblotting and immunohistochemistry | 3 months after bariatric surgery
Inflammation in adipose tissue using qRT-PCR, immunoblotting and immunohistochemistry | 6 months after bariatric surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Institut de recherches cliniques de Montréal, Montreal, Quebec, Canada